CLINICAL TRIAL: NCT04030572
Title: Pilot Study to Assess the Safety, Tolerability, and Feasibility of Administering Clonidine as a Pharmacological Challenge in Future Imaging Studies of Cerebrospinal Fluid Kinetics
Brief Title: Feasibility of Administering Clonidine as a Pharmacological Challenge in Imaging Studies
Acronym: a2a Agonist
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Not logistically feasible during the COVID pandemic
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-04020242
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Neuro-Degenerative Disease; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clonidine Pill (Experimental): One week period of clonidine, 0.1 mg tabs, one by mouth daily at bedtime
  Interventions: Drug: Clonidine Pill

INTERVENTIONS:
Drug: Clonidine Pill — 0.1 mg tabs, one by mouth daily at bedtime for one week
  Other Names: On-Drug

SUMMARY:
This will be a Phase 1, open label study of the pharmacokinetics (PK) and pharmacodynamics (PD) of clonidine, an alpha-2 adrenergic (a2a) agonist, in healthy volunteers. The primary aim is to show that the drug regimen is safe and reasonably well tolerated. The secondary aim is to demonstrate that safety can be monitored with home health devices.

DETAILED DESCRIPTION:
Subjects who screen in will participate in a drug-free lead-in period of one week duration. Then, the drug test article, clonidine HCl, 0.1 mg tabs, will be administered once daily by mouth at bedtime for one week. Steady-state PK will be measured on Day 8 post-drug with a single blood draw of 10 mL. This will be followed by a one week wash out period. During each of these three different one-week periods, sleep quality will be monitored nightly with a blue tooth and wireless enabled, wearable sleep tracker. Vital signs (VSs) will be monitored daily at home with a blue tooth and wireless enabled blood pressure machine. VSs and electrocardiograms (ECGs) will be measured before drug on Day (-7) and Day 1. Repeat measurements will be made during clinic visits on Day 2, Day 8, and Day 16.

The findings should show that there is, or is not, a PD effect produced by this rather low dose of drug administered for a relatively short period of time. Showing a PD effect at a safe and reasonably well tolerated dose would qualify this drug dosing regimen as a pharmacological challenge in future studies.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent.
* age 18-89
* Subjectively healthy and, in the opinion of the investigators, likely to be compliant with the drug regimen and the schedule of follow up visits.
* Normal hemodynamic function. Systolic blood pressure and pulse must be higher than 120 mmHg and 60 beats per minute while sitting. At the discretion of the investigators, athletic people who are in exceptionally robust condition may be enrolled if their systolic blood pressure and pulse are higher than 100 mmHg and 50 beats per minute while sitting.
* Unremarkable electrocardiograms with PR intervals of less than 200 mSec and QT intervals corrected with Fridericia's method (QTcF) of less than 440 mSec.
* No concurrent medications with the exception of p.r.n. NSAIDS, which must be discontinued one week prior to the lead-in period, and avoided for the next three weeks while on study (the one week lead-in period, one week on drug period, and one week washout period).
* Willing and able to refrain from abusing any recreational drugs, including marijuana because of its sleep effects, and drink less than one unit of alcoholic beverages per day starting one week prior to the lead-in period, and avoided for the next three weeks while on study (the one week lead-in period, one week on drug period, and one week washout period).
* Willing to refrain from donating blood while during the month of study.
* Willing to refrain from participating in any other research study that requires taking medication during the month of study.
* Willing to refrain from being vaccinated during the month of study.

Exclusion Criteria:

* History of allergy to clonidine.
* History of multiple hypersensitivity reactions, as indicated by allergies to multiple medications, foods, and seasonal pollen.
* History or physical examination suggestive of a condition, disorder, or disease that could represent a contra-indication to taking an antihypertensive. The relative contraindications to clonidine listed in the package insert under the section on precautions will be exclusionary in this study. They include subjects with coronary artery insufficiency syndromes, histories of myocardial infarction, cardiac conduction abnormalities, cerebrovascular disease, and chronic renal failure.
* Women who are pregnant or breast feeding will not be eligible to participate in the study, as clonidine is classified as a Class C risk to a fetus. (In fact, there is a safety signal in pregnant animal models that justifies exclusion, even if the signal is weak.)
* History or physical examination suggestive of a condition, disorder, or disease that could affect the adsorption, distribution, metabolism or excretion of the study drug.
* Positive urine toxicology screen for recreational drugs, other than cannabis.
* History of attention deficit hyperactivity disorder (ADHD) as a child or a residual disorder as an adult, because safety, tolerability, and patient acceptability have already been shown in these populations.
* Subjects may not be a member of a vulnerable population.
* May not have taken any controlled medications, including other study drugs, in the last 30 days or for 10 half-lives, whichever is longer.
* May not have donated blood in the 30 days prior to the start of the lead-in period.
* May not have participated in research administering drugs in the last 30 days.
* May not have been vaccinated in the 30 days prior to the start of the lead-in period.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events related to drug-induced changes in hemodynamic function. | Day 2 or Day 8 compared to Day (-7) through Day 1 during drug-free lead-in
  clinically significant drop in blood pressure or pulse

SECONDARY OUTCOMES:
Change in Total Sleep Duration | Day 2 and Day 8 on drug and Day 16 washout compared to Day (-7) through Day 1 during drug-free lead-in
  Time interval between falling asleep and waking up as estimated by a wearable sleep tracking device
Change in Deep Sleep Time | Day 2 and Day 8 on drug and Day 16 washout compared to Day (-7) through Day 1 during drug-free lead-in
  amount of time estimated to be in deep sleep versus light sleep by a wearable sleep tracking device

CONTACTS AND LOCATIONS:
Overall Officials: P. David Mozley, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified on-study data will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be made available within six months of last study visit or acceptance for publication, whichever comes first.
Access Criteria: Any reasonable request sent to dvm9029@med.cornell.edu